CLINICAL TRIAL: NCT01599052
Title: Social Cognition in Children Treated for a Brain Tumour: A Prospective Longitudinal Multi-Centre Study
Brief Title: Social Cognition in Children Treated for a Brain Tumour
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Radboud University Medical Center (Other); Universitaire Ziekenhuizen KU Leuven (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Dr. A. Kingma, Clinical Neuropsychologist, University Medical Center Groningen
Other Study IDs: 10.02.20-2010/0042; NL 31489.042.10 (Registry Identifier: CCMO)
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Social Behaviour; Brain Neoplasms; Cystic Fibrosis
Keywords: Social Cognition; Theory of Mind; Emotion Recognition; Social competence; Brain Tumour
MeSH Terms: conditions — Social Behavior; Brain Neoplasms; Cystic Fibrosis; Social Skills

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Brain Tumour Patients: Newly diagnosed brain tumour patients aged between 5 and 13 years
- Cystic Fibrosis patients: Patients diagnosed with Cystic Fibrosis aged between 5 and 13 years
- Healthy control group: Healthy children aged between 5 and 13 years

SUMMARY:
There is ample evidence that children treated for a brain tumour (BT) often develop deficits in social and emotional functioning. The investigators wish to examine the cause of these deficits, i.e. the underlying neuropsychological deficit(s). The aim is to study impairment and developmental delay in social cognition (and related cognitive functions) caused by brain damage in patients treated for a BT in childhood as compared to a reference group of chronically ill children. If we can identify the specific deficits these patients experience, neuropsychological treatment and guidance can be developed to give patients the most optimal chances to live as normal as possible, to improve their quality of life (QoL) and to prevent them from developing depression and anxiety. Eventually, an intervention programme could be developed based on our results, to improve social, vocational and emotional QoL.

DETAILED DESCRIPTION:
* Rationale: There is ample evidence that children treated for a brain tumour (BT) often develop deficits in social and emotional functioning. The investigators wish to examine the cause of these deficits, i.e. the underlying neuropsychological deficit(s). The following is expected:

  1. Children treated for a BT will perform worse than both healthy controls and patients with Cystic Fibrosis (CF) on measures of social cognition at Time 2 (3 years post diagnosis), but not at Time 1 (shortly after diagnosis, before neurotoxic treatment). The deterioration in performance will be influenced by the following adverse factors:

     1. History of cranial radiation therapy;
     2. Site of lesion in diencephalon;
     3. History of hydrocephalus and/or posterior fossa syndrome;
     4. Younger age at diagnosis.
  2. Parents and teachers will rate patients with a BT as being less socially competent and experiencing more internalizing problems than healthy controls and patients with CF at Time 2, but not at Time 1.
  3. Performance on tests of social cognition will be positively related to executive functions at Time 1 and 2.
  4. Performance on tests of social cognition will be positively related to parent and teacher reports of social competence and environmental biographic factors (parental education and occupation) at Time 1 and 2.
* Objective: To study impairment and developmental delay in social cognition (and related cognitive functions) caused by brain damage in patients treated for a BT in childhood as compared to a reference group of chronically ill children. The focus will be on the neurocognitive basis of such deficits.
* Study design: Comparative Non-randomised Prospective International Multi-Centre Study
* Study population: 49 Children treated for a BT aged 5-13 years, 32 children diagnosed with CF aged 5-13 years and 32 healthy controls aged 5-13 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5-13 years at first assessment (All groups)
* Newly diagnosed brain tumour patients that have not yet received adjuvant therapy (BT patients only)
* Stable medical condition (BT and CF patients only)

Exclusion Criteria:

* Diagnosed with a disorder of the autistic spectrum (Autism, Asperger's Syndrome or Pervasive Developmental Disorder not otherwise specified - All groups) that does not seem to be related to the tumour (BT patients only).
* History of other brain disease or neurological condition interfering with normal development (All groups).
* No native Dutch speaker (All groups)
* Severe sensory handicaps and/or behavioural problems interfering with reliable neuropsychological assessment (All groups)
* IQ below 70 (All groups)
* Poor prognosis and life expectancy less than 1 year (BT patients only)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Brain tumour (BT) patients will be recruited at paediatric oncology centres in Groningen (UMCG), Nijmegen (UMC St.Radboud), Amsterdam (VUmc) and Leuven (UZL).
  Cystic Fibrosis (CF) patients will be recruited at the department of paediatric lung diseases in Groningen (UMCG) and Nijmegen (UMC St. Radboud).
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2011-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Social cognitive performance | baseline and 3 years later
  Change in performance on tests of social cognition from time 1 (diagnosis) to time 2 (3 years later).

SECONDARY OUTCOMES:
Social-emotional competence | baseline and 3 years later
  Parent and Teacher reports of social and emotional functioning from time 1 (diagnosis) to time 2 (3 years later).
Influence of Biographical/Medical characteristics | up to 3 years later
  The influence of individual biographical and medical characteristics (age at diagnosis, histology, sex, tumor site, treatment) on change in performance on tests of social cognition from time 1 to time 2.

CONTACTS AND LOCATIONS:
Overall Officials: A Kingma, PhD, Principal Investigator — Unviersity Medical Centre
Locations (4):
- University Hospital Leuven, Leuven, Vlaams-Brabant, Belgium
- Netherlands (3):
  - University Medical Centre St. Radboud, Nijmegen, Gelderland
  - Vrije Universiteit Medical Centre, Amsterdam, North Holland
  - University Medical Centre Groningen, Groningen

REFERENCES:
- [Background] Kok TB, Post WJ, Tucha O, de Bont ES, Kamps WA, Kingma A. Social competence in children with brain disorders: a meta-analytic review. Neuropsychol Rev. 2014 Jun;24(2):219-35. doi: 10.1007/s11065-014-9256-7. Epub 2014 Mar 20. PMID 24648014
- [Background] Kok TB, Koerts J, Lemiere J, Post WJ, de Bont ESJM, Gidding C, Happe F, Jacobs S, Oostrom K, Schieving J, Tucha O, Kingma A. Social competence in newly diagnosed pediatric brain tumor patients. Pediatr Hematol Oncol. 2020 Feb;37(1):41-57. doi: 10.1080/08880018.2019.1682089. Epub 2019 Nov 4. PMID 31682775